CLINICAL TRIAL: NCT01487876
Title: A Randomized Controlled Trial of Dual-plasmid HBV DNA Vaccine Mediated by in Vivo Electroporation in Chronic Hepatitis B Patients Under Lamivudine Chemotherapy
Brief Title: Efficacy and Safety of Dual-plasmid Hepatitis B Virus DNA Vaccine in Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fuqiang Yang (Other)
Responsible Party: Sponsor-Investigator, Fuqiang Yang, Director of Department of Immunology and Biochemistry, Guangzhou 458 Hospital, The 458 Hospital of Chinese PLA
Organization: The 458 Hospital of Chinese PLA (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011005SW0101
Record Dates: First submitted 2011-09-22; First posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Hepatitis B
Keywords: DNA vaccine; HBV; Chronic hepatitis B (CHB); T-cell
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAM+DNA vaccine (Experimental): lamivudine (LAM) chemotherapy and DNA vaccine
  Interventions: Biological: HBV DNA vaccine
- LAM+Placebo (Placebo Comparator): Each volunteer received 4 injections of 4 mg placebo scheduled by a prime and 3 boosts at intervals of 4, 8, 12 weeks.
  lamivudine (LAM) chemotherapy and Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HBV DNA vaccine — HBV DNA vaccine means that each volunteer received 4 injections of 4 mg DNA vaccine scheduled by a prime and 3 boosts at intervals of 4, 8, 12 weeks.
  Arms: LAM+DNA vaccine
Other: Placebo — Placebo means the arm in which each volunteer received 4 injections of 4 mg placebo scheduled by a prime and 3 boosts at intervals of 4, 8, 12 weeks.
  Arms: LAM+Placebo

SUMMARY:
In order to study the immunotherapeutic effects of electroporation (EP)-mediated dual-plasmids Hepatitis B Virus DNA vaccine, the investigators plan to conduct a double-blind, randomized, placebo-controlled trial, approved by Chinese State Food and Drug Administration with written informed consent from each chronic hepatitis B (CHB) patients with baseline ALT more than 2 times the ULN, for whom antiviral treatment is indicated and who were under the simultaneous lamivudine (LAM) chemotherapy.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) affects approximately more than 350 million people worldwide, leading to a wide spectrum of clinical manifestations ranging from an asymptomatic carrier state to self-limited acute infection or fulminant hepatitis to chronic hepatitis with progression to cirrhosis and hepatocellular carcinoma and poses a serious public health problem in endemic counties like China. Current available therapeutic remedies such as interferons and nucleotide/nucleoside analogues are far from satisfactory, for their therapeutic efficacies are limited by the high economic cost with the less tolerable adverse effects or the lack of viral eradicative effect for its long term control of the virus in most of the patients. Viral persistence has been associated with a defect in the development of HBV-specific cellular immunity. Strategies to boost or to broaden the weak virus-specific T-cell response of patients with chronic hepatitis B have been proposed as a means of curing this persistent infection. HBV envelope- and nucleocapsid-based vaccines, new formulations for recombinant vaccines and DNA-based vaccines are currently being assessed in clinical trials, among which DNA vaccine represents a promising immunotherapeutic approach that can induce T-cell mediated antigen specific immunity, owing to its de novo intracellular antigenic protein expression and synthesis.

In clinical trials, although HBV DNA vaccination developed protective antibody responses and antigen-specific CD8 T cells in healthy hepatitis-naive human volunteers, the detectable HBV-specific IFN-γ secreting T cells and decreased serum HBV DNA levels only in some chronic HBV carriers vaccinated with HBV PreS2/S DNA vaccine were limited. One resolution for the main obstacles of the new technique development is to enhance the transfection efficiency of plasmids into host cells; the other is to improve the immunogenicity of DNA vaccine by driving the naïve T cell responses towards the Th1 profile. To tackle the first problem of low transfection rate of DNA vaccine, the investigators had applied the in vivo electroporation (EP) for potency enhancement of HBV DNA vaccine, which dramatically improved the host cell transfection of the plasmids and enabled the DNA vaccine the investigators prepared to elicit both humoral and cellular immune responses in the large body weight animals like rabbit and nonhuman primates. In order to achieve the second goal of immunogenicity improvement of HBV DNA vaccine for its therapeutic usage, the investigators had designed and constructed the Th1 type cytokines (interleukin-2 and interferon-γ) fusion protein expression gene plasmids (pFP), in attempt to direct Th1 bias in favor of cellular immunity augment when being used in combination with HBV DNA vaccine. Both tactics in the form of the dual-plasmids DNA vaccination mediated by EP have been investigated to be safe and efficient to improve the transfection and enhance the immunogenicity of DNA vaccine to the host in both animal models and in phase I,II trials of healthy volunteers and CHB patients.

In order to study the immunotherapeutic effects of EP-mediated dual-plasmids HBV DNA vaccine, the investigators plan to conduct a clinical trial, approved by Chinese State Food and Drug Administration (license number: 2006L03542) with written informed consent from each patient. The trial is a double-blind, randomized, placebo-controlled one in CHB patients with baseline ALT more than 2 times the ULN, for whom antiviral treatment is indicated and who were under the simultaneous lamivudine (LAM) chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years with either sex;
2. HBV serology meet the following criteria:

   * HBsAg-positive lasting for at least 6 months at the time of screening;
   * HBeAg-positive at the time of screening;
   * Serum HBV DNA≥1.0×10E5 copies/ml at the time of screening
3. 80U/L<ALT<400U/L;
4. TBIL<40μmol/L;
5. No YMDD mutation of the HBV drug resistance gene
6. Subjects agree not to participate in any other clinical trial or take any other anti-HBV therapeutics during the study;
7. Subjects understand and sign the ICF which approved by EC, and are able to comply with the study procedures and complete the study.

Exclusion Criteria:

1. Was suspected with HCC by the following evidence:

   * B-Ultrasound or imaging which shows occupying lesions;
   * Continuingly elevating serum AFP level even if the B-Ultrasound is normal;
   * AFP >100ng/ml;
2. With acute hepatic decompensation caused by liver disease aggravation or with clinical symptoms of decompensated liver disease at baseline;
3. Serum Cr≥1.5mg/dl (≥130μmol/l) at the time of screening;
4. Serum amylase > two-fold of the upper limit of the normal reference value;
5. Hb (male<100g/ L, female<90g/L), WBC<3.5×10E9/L,PLT<60×10E9/L (except hypersplenism and cirrhosis);
6. Co-infection with HCV (anti-HCV positive), HIV and anti-HAV IgM positive, anti-HDV IgM positive, anti-HEV IgM positive, anti-CMV IgM positive and autoimmune hepatitis (e.g. antinuclear antibody titer>1:160 ) or other active liver disease caused by known or unknown factors;
7. Any other serious disease or active diseases other than hepatitis B that are considered by investigators to be potential factors that may interfere with the therapy, assessment or compliance with the protocol, including any uncontrolled diseases with clinical significance, e.g. kidney, heart, lung, blood vessel, neurogenic, digestive system and metabolic diseases (diabetes, hyperthyroidism, adrenal gland diseases), autoimmune dysfunctions, and tumors, etc;
8. History of alcohol or drug abuse that is considered by investigators that could affect subject's compliance with the protocol or could influence the result of the analysis;
9. Pregnant or breast-feeding female subjects, or those who plan to be pregnant during the course of the study or male subjects' companions who plan to be pregnant during the course of the study;
10. Having used immunosuppressive agents, immunomodulators (thymosin), cytotoxic drugs within 6 months or transaminase-decreasing drugs within one month prior to the initiation of this study;
11. Having used anti-HBV drugs (Lamivudine, interferon, adefovir, entecavir, or sebivo, etc.) within 6 months prior to the initiation of this study;
12. Had or planning to have liver transplantation;
13. Having received experimental drug treatment from any other study within 3 months prior to the screening;
14. Allergic to nucleoside drugs or nucleoside analogues;
15. Not agreeing to the study protocol or any other factors considered not eligible for this study by investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
HBV DNA suppression | Before and after DNA vaccine injection: weeks 0, 60.
  Suppression of HBV DNA was defined as the >2 log10 decrease of viral load from baseline level.
Loss of HBeAg | Weeks 0, 48.
  HBeAg serum titer was dropped to the detection limit by quantitative determination.
Appearance of Anti-HBe | At weeks 0,48.

SECONDARY OUTCOMES:
HBeAg seroconversion rate | At weeks 0, 12, 24, 48, 72.
  loss of HBeAg, or presence of anti-HBe antibody
The occurrence of YMDD mutants | At weeks 0, 48, 72.
  Tyrosine-methionine-aspartate-aspartae (YMDD) mutants were evaluated by means of polymerase chain reaction-restricted fragment length polymorphism (PCR-RFLP) and PCR-Sequencing (Invitrogen Ltd. Shanghai,China), at baseline, week 48 and 72. The amino acid (AA) mutations were identified by comparing HBV RT sequences with the genotype-matched consensus sequence generated based on the HBV sequences obtained from genbank. A mutation type was referred to the replacement of the consensus AA of the corresponding genotype with a novel one.
Viral breakthrough rate | At weeks 0, 12, 24, 40, 48, 56, 60, 64, 72.
  On the basis of present Guideline for Management of chronic hepatitis B (CHB), the virologic breakthrough (VBT) was defined as >1 log copies increase in HBV DNA from nadir after an initial virologic response or HBV DNA could be detected again after the previous report of "under the detection limit".
HBV Ag specific T cell immunity | At weeks 0, 12, 24, 36, 52, 72.
  The enzyme-linked immunosorbent spot (ELISPOT) assay was performed according to the manufacture's protocol in the human IFN-g ELISPOT Set (BD Biosciences, San Diego, CA, USA). The ELISPOT assay for enumeration of antigen-specific IFN-γ-secreting cells (spot forming cells, SFCs) was performed according to the manufacturer's instructions . The number of IFN-γ spots was counted by AID Elispot reader system (AID, Germany). Data are expressed as the mean SFCs/106 PBMC.
  Detection of HBV-specific cytotoxic T lymphocyte (CTL) was performed by using flow cytometry (FACS) Calibur (BD Biosciences).

CONTACTS AND LOCATIONS:
Locations (1):
- Guiqiang Wang, Beijing, Bejing, China